CLINICAL TRIAL: NCT05411484
Title: Self-controlled, Single-site Trial Investigation of Laser Assisted Drug Delivery of NanoDOX®
Brief Title: Investigation of Laser Assisted Drug Delivery of NanoDOX®
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NanoSHIFT LLC (Industry)
Responsible Party: Principal Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001117
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Wounds and Injury
Keywords: WOUND; DRUG-DELIVERY
MeSH Terms: conditions — Wounds and Injuries | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Self-controlled single-site study of healthy subjects receiving an ablative fractional CO2 laser procedure followed by topical application of NanoDOX® Hydrogel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pilot Arm (Experimental): Self-controlled 12 healthy subjects receiving an ablative fractional CO2 laser procedure followed by topical application of NanoDOX® Hydrogel
  Interventions: Drug: NanoDOX® Hydrogel; Device: CO2 Ablative Fractional Laser

INTERVENTIONS:
Drug: NanoDOX® Hydrogel — NanoDOX® Hydrogel (Doxycycline Monohydrate USP) will be applied on the areas of the skin previously treated by the Co2 Ablative Fractional Laser and also on a small non treated area of the subject's skin
  Other Names: Doxycycline application
Device: CO2 Ablative Fractional Laser — CO2 Ablative Fractional Laser will be applied to healthy skin areas
  Other Names: laser treatment

SUMMARY:
This is a self-controlled single-site study of healthy subjects receiving an ablative fractional CO2 (carbon dioxide) laser procedure followed by topical application of NanoDOX® Hydrogel (1% doxycycline). The study includes skin biopsies to evaluate the effects of NanoDOX® Doxycycline Monohydrate Gel on wound healing after the ablative laser procedure. Study subjects will be asked to do 2 visits of 4 hours in total over approximately 1 week. An optional third visit will take place approximately 6 weeks after Visit 1. In this study, 20 subjects are expected to enroll with a goal of 12 healthy subjects to enroll and complete the study.

DETAILED DESCRIPTION:
Effective topical delivery of any pharmaceutical agent requires small molecule drugs to penetrate the epidermis, yet the absorption of topical products through the epidermis is limited.

In this study, the investigators are looking for healthy volunteers who are eligible to help us to determine the safety and efficacy of ablative fractional laser therapy combined with NanoDOX. The investigators are doing the research to evaluate drug delivery of topical NanoDOX® Hydrogel following ablative fractional CO2 laser treatment and our secondary objective is to evaluate the efficacy of NanoDOX® for wound healing.

Subjects will have a screening visit to determine eligibility, 2 study visits when they will receive CO2 ablative fractional laser treatment, NanoDOX® Hydrogel application, and skin biopsies, and 1 optional study visit for wound healing assessment. Laser procedure will happen only during visit 1, visit 2 will happen 2 days after visit 1, and visit 3 will happen approximately 6 weeks after visit 1. In total, 7 skin biopsies will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
* Subject must be able to read and understand English;
* Any gender and any Fitzpatrick skin type;
* Age equal to or greater than 18 years old;
* Willing to sun protect treated area (sunscreen or cover the area with clothes) for the duration of enrollment in the study and 1 year after treatment.
* Subjects must be willing to undergo skin biopsies

Exclusion Criteria:

* Participation in another investigational drug or device clinical trial in the past 30 days;
* Are pregnant or lactating;
* History of allergic reaction to topical or local anesthesia;
* History of allergic reaction to Doxycycline or other tetracyclines;
* Regular intake of high doses of anti-inflammatory drugs (aspirin >81 mg/day, ibuprofen, corticosteroids, etc.) , immunosuppressive drugs or biologics;
* Clinically significant abnormal findings or conditions which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study;
* Laser treatment in past six months; History of poor wound healing;
* History of keloids; History of extreme photosensitivity;
* History of severe hyperpigmentation; History of tattoos on thighs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Skin drug uptake | 3 days
  The depth of drug uptake will be measured by histology analysis. To determine if ablative fractional laser therapy combined with NanoDOX® topical drug improves the depth of drug uptake, fluorescence microscopy will be used to measure the concentration of the drug inside the skin by the amount of fluorescence created by the drug will be quantified.

SECONDARY OUTCOMES:
Wound healing | 6 weeks
  Biopsied areas will not be sutured, so wound healing will be evaluated by clinical assessment; the investigators will assess the wounds on the untreated and treated areas with NanoDOX® Hydrogel after ablative fractional laser.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials And Outcome, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Waibel JS, Wulkan AJ, Shumaker PR. Treatment of hypertrophic scars using laser and laser assisted corticosteroid delivery. Lasers Surg Med. 2013 Mar;45(3):135-40. doi: 10.1002/lsm.22120. Epub 2013 Mar 4. PMID 23460557
- [Background] Alegre-Sanchez A, Jimenez-Gomez N, Boixeda P. Laser-Assisted Drug Delivery. Actas Dermosifiliogr (Engl Ed). 2018 Dec;109(10):858-867. doi: 10.1016/j.ad.2018.07.008. Epub 2018 Sep 25. English, Spanish. PMID 30266385
- [Background] Qu L, Liu A, Zhou L, He C, Grossman PH, Moy RL, Mi QS, Ozog D. Clinical and molecular effects on mature burn scars after treatment with a fractional CO(2) laser. Lasers Surg Med. 2012 Sep;44(7):517-24. doi: 10.1002/lsm.22055. Epub 2012 Jul 31. PMID 22907286
- [Background] Waibel JS, Rudnick A, Shagalov DR, Nicolazzo DM. Update of Ablative Fractionated Lasers to Enhance Cutaneous Topical Drug Delivery. Adv Ther. 2017 Aug;34(8):1840-1849. doi: 10.1007/s12325-017-0516-9. Epub 2017 Jul 7. PMID 28687935
- [Background] Benzaquen M, Collet-Villette AM, Delaporte E. Combined treatment of hypertrophic and keloid scars with intralesional injection of corticosteroids and laser-assisted corticosteroid delivery. Dermatol Ther. 2019 Nov;32(6):e13126. doi: 10.1111/dth.13126. Epub 2019 Nov 6. No abstract available. PMID 31628774
- [Background] Moore AL, desJardins-Park HE, Duoto BA, Mascharak S, Murphy MP, Irizarry DM, Foster DS, Jones RE, Barnes LA, Marshall CD, Ransom RC, Wernig G, Longaker MT. Doxycycline Reduces Scar Thickness and Improves Collagen Architecture. Ann Surg. 2020 Jul;272(1):183-193. doi: 10.1097/SLA.0000000000003172. PMID 30585822